CLINICAL TRIAL: NCT06573008
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Phase III Clinical Study on the Safety and Efficacy of GP681 Tablets in Patients With Influenza at High Risk of Influenza Complications
Brief Title: Study of GP681 Tablets Compared With Placebo in Patients With Influenza at High Risk of Influenza Complications
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GP681-202402
Record Dates: First submitted 2024-08-18; First posted 2024-08-27 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Influenza, Human
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GP681 tablet 40mg (Experimental): Patients in the GP681 tablet 40mg group will receive a single oral dose of GP681 tablet 40mg.
  Interventions: Drug: GP681 40mg
- Placebo group (Placebo Comparator): Patients in the Placebo group will receive a single oral dose of GP681 Simulant 40mg.
  Interventions: Drug: GP681 Simulant

INTERVENTIONS:
Drug: GP681 40mg — 2 x 20mg tablets taken orally
  Arms: GP681 tablet 40mg
Drug: GP681 Simulant — Placebo tablets matching GP681 40mg
  Arms: Placebo group

SUMMARY:
This study will evaluate the efficacy, safety, and population pharmacokinetics of a single, oral dose of GP681 compared with placebo in patients aged 12 and older With Influenza at High Risk of Influenza Complications.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients aged ≥12 years at the time of signing the informed consent form.
2. Patients with a diagnosis of influenza confirmed by all of the following:

   * Positive throat or nose swab by rapid influenza antigen test (RAT) (where rapid influenza virus nucleic acid test or other rapid molecular diagnostic methods are also acceptable);

     * Fever (axillary temperature ≥37.3℃) in the predose examinations or > 4 hours after dosing of antipyretics if they were taken;

       * At least one of the following systemic symptoms and respiratory symptoms respectively associated with influenza are present with a severity of moderate or greater:

   Systemic symptoms: headache, fever or chills, muscle or joint aches, fatigue; Respiratory system symptoms: cough, sore throat, nasal congestion.
3. The time interval between the onset of symptoms and random enrollment is 48 hours or less. The onset of symptoms is defined as either:

   1. Time of the first increase in body temperature (axillary temperature ≥37.3℃)
   2. Time when the patient experiences at least 1 new general or respiratory symptom related to influenza
4. Referring to the standards of the Centers for Disease Control and Prevention (CDC) in the United States and the definition of high-risk populations for influenza complications in the "Expert Consensus on Diagnosis and Treatment of Influenza in Adults in the Emergency Department (2022 Edition)", that is, if at least one of the following criteria is met, the patient will be considered at high risk of influenza complications:

   1. Asthma or chronic lung diseases [such as chronic obstructive pulmonary disease (COPD), cystic fibrosis, chronic bronchitis, bronchiectasis, emphysema, chronic interstitial pneumonia, etc.];
   2. Endocrine disorders (including diabetes);
   3. Residents of long-term care institutions (such as nursing homes);
   4. Immune system impairment (including patients receiving chronic systemic corticosteroid treatment of ≤20mg/d prednisone or an equivalent dose);
   5. Neurological and neurodevelopmental disorders (including brain, spinal cord, peripheral nerve and muscle diseases, such as cerebral palsy, epilepsy (episodic disorders), stroke, muscular dystrophy or spinal cord injury);
   6. Heart diseases (such as congenital heart disease, congestive heart failure, or coronary artery disease), but not including hypertension without any other cardiac-related symptoms;
   7. Patients aged ≥65 years;
   8. Blood system diseases (such as sickle cell disease);
   9. Metabolic system diseases (such as hereditary metabolic diseases and mitochondrial diseases);
   10. Liver diseases (such as chronic hepatitis B, chronic hepatitis C, non-alcoholic steatohepatitis);
   11. Kidney diseases (estimated glomerular filtration rate eGFR ≥ 30 mL/min/1.73m2 by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula);
   12. Obese patients (BMI ≥ 30 kg/m2);
   13. Female patients within 2 weeks postpartum and not breastfeeding.
5. Subjects of child-bearing potential who agree to use a highly effective method of contraception for 1 month after drug withdrawal.
6. Subjects and/or their guardian who are willing to provide written informed consent and consent to participate in the study, able to understand the study and comply with all study procedures, including patient health diary records.

Exclusion Criteria:

1. History of allergic reactions attributed to GP681,Acetaminophen, bromohexine hydrochloride or any of the ingredients of its formulation.
2. Known history of dysphagia or any gastrointestinal disease that affects drug absorption (including but not limited to chronic diarrhea, inflammatory bowel disease, tuberculosis of the intestines, gastrinoma, short bowel syndrome, postoperative gastrectomy, etc.);
3. Screening patients who, in the opinion of the investigator, require hospitalization due to severe influenza virus infection;.
4. Screening patients who, at the time of screening, are clinically diagnosed with bacterial or other viral infections requiring systemic antibacterial or antiviral treatment;
5. Cancer patients who are currently receiving or have received chemotherapy or radiation therapy within the past year (excluding non-melanoma skin cancer and thyroid cancer)
6. Known HIV-infected patients;
7. Organ or bone marrow transplant recipients;
8. Patients who are currently receiving >20mg/d of prednisone or equivalent chronic systemic corticosteroid therapy;
9. Patients who have used anti-influenza virus drugs (including neuraminidase inhibitors, hemagglutinin inhibitors, and M2 ion channel blockers, such as oseltamivir, zanamivir, palivizumab, favipiravir, abidol, marabolexavir, amantadine or rimantadine or other anti-influenza virus drugs approved by NMPA) within the past 2 weeks or who have received influenza vaccination within the past 6 months;
10. Exclusion of participants who have received clinical research or screening within the past 30 days for any indication with a trial drug or device, or who have received clinical research for a monoclonal antibody drug for viral diseases within the past year;
11. Known to have had a previous history of severe liver function impairment such as cirrhosis with ascites, hepatic encephalopathy, or a history of upper gastrointestinal bleeding;
12. Estimated glomerular filtration rate (eGFR) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula <30mL/min/1.73m2 at the time of screening;
13. Individuals with a history of alcohol abuse or substance abuse (more than 14 units of alcohol per week, 1 unit of alcohol = 360 mL of beer or 45 mL of spirits with an alcohol content of 40% or 150 mL of wine with an alcohol content of 12%);
14. Adult reproductive-age females who are pregnant or breastfeeding or who have a positive pregnancy test. Women who are infertile (i.e., women who have had a hysterectomy, bilateral oophorectomy, or tubal ligation for medical reasons or who are postmenopausal - defined as age > 50 years and menopause has occurred for at least 2 years) do not need a pregnancy test;
15. Patients who, in the opinion of the Investigator, may not be qualified or suitable for the study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 328 (Estimated)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Time to alleviation of influenza symptoms | up to Day 15
  Participants assessed the severity of seven influenza-associated symptoms (cough, sore throat, headache, nasal congestion, feverishness or chills, muscle or joint pain, and fatigue) on a 4-point scale (with 0 indicating no symptoms, 1 mild symptoms, 2 moderate symptoms, and 3 severe symptoms).
  Defined as the time from the start of treatment until the patient's body temperature returns to normal and all 7 flu symptoms (cough, sore throat, headache, nasal congestion, fever or chills, muscle or joint pain, fatigue) have alleviated (scoring 0 or 1 point), maintained, or improved, as defined below, for at duration of at least 21.5 hours.
  Preexisting symptoms (cough, fatigue, or muscle/joint pain that existed prior to influenza) that were worse at baseline must have improved at least 1 point from baseline Preexisting symptoms not worse at baseline must have maintained baseline severity New symptoms must have alleviated, defined as a symptom score of none (0) or mild (1).

SECONDARY OUTCOMES:
Change From Baseline in Virus RNA (Q-PCR) at Each Time Point | Day 2, Day3, Day5, Day7
  Nasopharyngeal swabs were obtained for viral quantitation.
Percentage of Participants With Positive Influenza Virus RNA by Q-PCR at Each Time Point | Day 2, Day3, Day5, Day7
  The percentage of patients positive for virus RNA by RT-PCR.
Area Under the Concentration (AUC) of virus RNA by Q-PCR and AUC of virus titer | Up to Day 7
  AUC of the viral load by RT-PCR and AUC of viral titer measured from baseline to Day 7
Change in the total score of 7 influenza symptoms | Up to Day15
  The composite symptom score is the total score of the 7 influenza symptoms(Sum of symptom scores) as assessed by the participant, and ranges from 0 to 21.
Time to Cessation of Viral Shedding Determined by Virus Titer | up to Day7
  Defined as the time between the initiation of the study treatment and first time when the virus titer was below the limit of detection.
Time to alleviation of each influenza symptom. | Up to Day15
  Defined as the time from the start of the study treatment to the start of the time when the individual symptom was assessed by the participant as have alleviated (scoring 0 or 1 point), maintained, or improved , for at duration of at least 21.5 hours.
Time to Alleviation of the Three Respiratory Symptoms in Participants | Up to Day15
  Defined as the time from the start of study treatment to the time when all 3 respiratory symptoms (cough, sore throat, and nasal congestion) were alleviated, maintained, or improved, as defined below, for a duration of at least 21.5 hours.
Time to Alleviation of the Four Systemic Symptoms in Participants | Up to Day15
  Defined as the time between the initiation of study treatment to the time when all 4 systemic symptoms (headache, feverishness or chills, muscle or joint pain, and fatigue) were alleviated, maintained, or improved, for a duration of at least 21.5 hours.
Percentage of Participants Reporting Normal Temperature at Each Time Point | 12h, 24h,48h,72h,96h,120h,144h,168h
  Defined as the percentage of patients whose axillary temperature dropped to less than 37.3ºC after the initiation of study treatment
Time to Resolution of Fever | Up to Day15
  Defined as the time between the initiation of the study treatment and the resolution of fever. The resolution of fever was defined as the time when the participant's self-measured axillary temperature became less than 37.3ºC and was maintained at less than 37.3ºC for a duration of at least 21.5 hours.
Incidence of influenza-related complications | Up to Day15
  Defined as the percentage of subjects in the analysis population who experience each influenza-related complication (hospitalization, death, sinusitis, bronchitis, otitis media, and pneumonia) as an adverse event after the initiation of the study treatment.
Proportion of patients and frequency in combination use of acetaminophen. | Up to Day15
  The proportion of patients who use acetaminophen in the duration of the study
The percentage of participants who received systemic antibiotics. | Up to Day15
  The proportion of patients receiving systemic antibiotic therapy after treatment initiation.
The percentage of participants with secondary influenza infections after enrollment | Up to Day15
  Defined as the percentage of subjects who develop secondary influenza infections after treatment initiation in the study population as an adverse event after the initiation of the study treatment
Time to Return to Preinfluenza Health Status | Up to Day15
  Defined as the participant's pre-influenza daily activity score from the start of treatment until the participant's recovery to influenza. Subjects whose baseline self-reported daily activity score was higher than or equal to the pre-influenza score were excluded from the analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- The people's Hospital of Chizhou, Chizhou, China

IPD SHARING:
Plan to Share IPD: No